CLINICAL TRIAL: NCT06008353
Title: A Real-World Assessment of the Demographic, Clinical Characteristics and Outcomes of a Brazilian Cohort of Previously Untreated Extensive Stage-Small Cell Lung Cancer Receiving Durvalumab Combined With Platinum-Etoposide in (ES-SCLC) in Brazil
Acronym: EDUR-BRA
Status: Active, not recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D4191R00053; D4191R00053 (Other Grant/Funding Number: AstraZeneca)
Record Dates: First submitted 2023-03-07; First posted 2023-08-23 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Extensive-stage Small-cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult patients newly diagnosed with ES-SCLC: The study will include consecutive adult patients newly diagnosed with ES-SCLC (patients with the recurrent limited stage disease are also eligible).
  Interventions: Other: Observational study

INTERVENTIONS:
Other: Observational study — This is an observational study; patients will not be exposed to clinical interventions different from those belonging to the standard of care.

SUMMARY:
The central objective of this study is to characterize the demographic of an ES-SCLC Brazilian cohort treated with durvalumab. Secondarily, to assess the outcomes of durvalumab-based regimens in 1L treatment of ES-SCLC Brazilian patients from the private health care setting.

ELIGIBILITY:
Inclusion Criteria:

* Have a documented diagnosis of ES-SCLC (newly diagnosed patients, as well as limited stage relapsed patients, are eligible);
* Have been treated with a durvalumab-based regimen for 1L ES-SCLC in the past (retrospective) OR is currently being treated with a durvalumab-based regimen for 1L ES-SCLC (prospective);
* Male or female adult patients ≥ 18 years of age (as per local Durvalumab approved label);
* Provision of consent in a signed informed consent form (ICF) (allowing for data to be captured from existing medical records). If the patient´s data is entirely retrospective (i.e., the patient already presented progression, death, or completed 18 months of durvalumab-based treatment), the ICF may be waived, as decided by the local ethics committee.

Exclusion Criteria:

* Since the study is observational, there are no Exclusion Criteria. If the patient meets all the Inclusion Criteria, he/she will be eligible for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male or female patients (aged 18 years or older) with histologically- or cytologically-documented ES-SCLC receiving a durvalumab-based regimen as a first-line treatment.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-01-18 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Demographic Characteristics of the Cohort | Baseline.
  This measure encompasses relevant demographic information of the patients included in the cohort, including median age at diagnosis, gender distribution, smoking history, and World Health Organization Performance Status (WHO PS) score. These details will provide a comprehensive understanding of the patient profile within the cohort.
Clinical Characteristics of the Cohort | Baseline.
  This measure encompasses relevant clinical information of the patients included in the cohort, including presence of hepatic and cerebral metastases, type of platinum used in first-line (1L) treatment, and diagnostic stage (III vs. IV) of CPPC-EE. These details will provide a comprehensive understanding of the patient profile within the cohort.
Comparison of Demographic and Clinical Characteristics between Recurrent and Newly Diagnosed CPPC-EE Patients | During the cohort follow-up, an average of 24 months, starting from diagnosis.
  This measure focuses on comparing patients with recurrent CPPC-EE and those newly diagnosed. The incidence of disease recurrence and distinct demographic and clinical characteristics between these groups, such as age, gender, smoking history, World Health Organization Performance Status (WHO PS) score, presence of hepatic and cerebral metastases, type of platinum used in first-line (1L) treatment, and diagnostic stage, will be analyzed and reported. This will allow for a deeper understanding of differences between recurrent and newly diagnosed patients.

CONTACTS AND LOCATIONS:
Overall Officials: Mauro Zukin, Principal Investigator — Latin American Cooperative Oncology Group
Locations (5):
- Brazil (5):
  - ÉTICA Clínica AMO - Assistência Multidisciplinar em Oncologia, Salvador, Estado de Bahia
  - Oncologia D'Or Unidade Esperança Pernambuco, Recife, Pernambuco
  - Instituto D'Or de Pesquisa e Ensino RJ, Rio de Janeiro
  - BP - A Beneficência Portuguesa de São Paulo, São Paulo
  - A.C. Camargo Cancer Center, São Paulo

IPD SHARING:
Plan to Share IPD: No